CLINICAL TRIAL: NCT04569708
Title: Auditory Stimulation Effect on Spindles and Sleep Dependent Learning in Rolandic Epilepsy
Brief Title: Sleep Spindles and Memory in Rolandic Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Catherine Chu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020P002668; 1R01NS115868-01 (NIH)
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Rolandic Epilepsy; Rolandic Epilepsy, Benign; Centrotemporal Epilepsy; Centrotemporal; EEG Spikes, Epilepsy of Childhood; Epilepsy; Seizure; Epilepsy
MeSH Terms: conditions — Epilepsy, Rolandic; Epilepsy | interventions — Acoustic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children and adolescents with epilepsy and controls (Experimental): Closed loop auditory stimulation during nap
  Interventions: Other: Auditory stimulation

INTERVENTIONS:
Other: Auditory stimulation — Quiet auditory stimulation timed with sleep physiology

SUMMARY:
The investigators are recruiting children with Rolandic epilepsy and children without epilepsy (aged 4 years old and above) for a non-invasive brain imaging study using Magnetic Resonance Imaging (MRI), Magnetoencephalography/Electroencephalography (MEG/EEG), and experimental tasks. The investigators hope to determine the brain circuits and brain rhythms affected in these children and ultimately identify new treatment options for childhood epilepsy patients.

DETAILED DESCRIPTION:
This is a prospective study of epilepsy biomarkers in a total of 100 subjects of ages 4-18. Participants will spend about 5 hours at the Massachusetts General Hospital (MGH) Athinoula A. Martinos Center for Biomedical Imaging. They will undergo training on a memory task concurrent with EEG/MEG recordings. During the EEG, subjects will wear headphones that will deliver a quiet pink noise stimulus intermittently during a nap. The auditory stimulus will be calibrated in volume to not cause arousals. After napping, subjects will undergo cognitive testing and memory task testing.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 4-18 years
2. Diagnosed with childhood epilepsy with centrotemporal spikes (CECTS) or Rolandic epilepsy by child neurologist
3. Has EEG with sleep activated centrotemporal spikes
4. Has had at least 1 focal motor or generalized seizure

Exclusion Criteria:

1. Has abnormal brain MRI
2. Has other unrelated neurological disease
3. Unable to have an MRI/MEG

   1. Claustrophobic
   2. History of frequent vomiting
   3. Permanent metal in body, braces
   4. Over MRI weight limit: 350lbs

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Spindle Density | 1-5 hours
  Spindle count per minute during non-rapid eye movement (NREM) sleep
Memory performance | 1-5 hours
  Percent improvement in memory task performance

OTHER OUTCOMES:
Spindle-slow oscillation coupling | 1-5 hours
  Cross frequency coupling

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Athinoula A. Martinos Center Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Derivative data will be shared with appropriate IRB approval per publication requirements
Supporting Information: Analytic Code
Time Frame: 2020 - 2030
Access Criteria: In accordance with IRB approval